CLINICAL TRIAL: NCT07054788
Title: Effect of Kinesiotaping on Lower Limb Kinematics and Functional Related Outcomes Among Female Athletes With Chronic Lateral Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelaziz Abdel Moneim Elnakee, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mahmoud-005551
Record Dates: First submitted 2025-06-28; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Kinesiotapping; Kinematics; Athletes Foot; Chronic Ankle Instability
MeSH Terms: conditions — Tinea Pedis | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy with Kinesiology tape (Experimental): This group involves fifty-five participants and will receive kinesiology tape with mobilization with movement and calf muscle flexibility exercises. 3 sessions per week for 2 weeks.
  Interventions: Other: Flexibility Exercise; Other: Mulligan mobilization with movement; Other: Kinesiology Taping
- Exercise therapy with placebo tap (Active Comparator): This group involves fifty-five participants and will receive mobilization with movement and calf muscle flexibility exercises and placebo tape. 3 sessions per week for 2 weeks.
  Interventions: Other: Flexibility Exercise; Other: Mulligan mobilization with movement; Other: Placebo tape

INTERVENTIONS:
Other: Flexibility Exercise — Participants will perform calf muscle stretching exercises. The participant will be asked to keep the knee of the stretched leg straight with the heel flat on the ground, slightly bend the front knee, and push the hips toward a wall.
  The exercise will be done in 2 sets of 3 repetitions, every repetition for 30 seconds and a ten-second rest, with a one-minute rest between sets
Other: Mulligan mobilization with movement — The Mulligan mobilization techniques involve talar glide and fibular glide. Talar glide involves manually stabilizing the patient's talus and leg with anteroposterior direction pressure, while fibular glide involves a pain-free sustained anterior to posterior, slightly superior, and lateral glide of the distal fibula. The patient is then asked to plantar-flex, invert the foot, and perform overpressure. The technique is performed during ankle dorsiflexion in a closed kinetic chain.
Other: Kinesiology Taping — The length of tape is calculated using a formula: B = A + (XA ∗ 0.35), where "A" is the tape's length, "X" is the pretension, "0.35" is the 35% tension, and "B" is the muscle's length from origin to insertion. In this study, 50% pretension was used, and "A" was added to the tails. Fibular taping is applied immediately after the MWM to improve positional alignment, wrapping around the distal tibia and applying Mueller tape in the same direction. Talar taping involves wrapping Mueller tape from the talus downward and posterior to the calcaneus while holding the ankle in slight dorsiflexion.
  Arms: Exercise therapy with Kinesiology tape
Other: Placebo tape — The formula for cutting tape length is B = A + (XA ∗ 0.35), where "A" represents the tape's length, "X" is the pretension, "0.35" is the 35% tension, and "B" is the muscle's length from origin to insertion. In this study, 50% pretension was used, and "A" was added to the tails' length. The tape application involves two steps: from below the medial calcaneus to the medial aspect of the lower leg, and from below the lateral malleolus to the lateral aspect.
  Arms: Exercise therapy with placebo tap

SUMMARY:
The current study aims to measure the effect of adding kinesiology tape to ankle mobilization with movement with calf muscles flexibility exercise on dorsiflexion range of motion, dynamic balance, lower limb kinematics, and self-reported physical function versus mobilization with movement, calf muscles flexibility exercise, and placebo kinesiotapping in female basketball players with unilateral chronic lateral ankle instability

DETAILED DESCRIPTION:
Chronic ankle instability affects up to 70% of individuals with lateral ankle sprain, causing pain, recurrent sprains, and instability. This condition significantly impacts physical and financial welfare, necessitating effective treatment techniques. Ankle injuries are common in healthy, active individuals, affecting women more frequently than men. These injuries can cost healthcare systems around the United States dollars 6.2 billion in high school athletes in the United States and euro 208 million in the Netherlands annually. Most rehabilitation protocols focus on isolated interventions, neglecting the potential benefits of combined strategies. This study contributes to evidence-based practice by adding to existing knowledge on chronic ankle instability rehabilitation practices and supporting healthcare professionals in implementing effective treatment plans. Combined intervention strategies may enhance dorsiflexion range of motion, lower limb kinematics, ankle stability, postural control, and athletic performance, reducing time away from sports.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-24 years.
2. chronic ankle instability group has a history of unilateral ankle inversion injury since at least one year before the study onset
3. A period of restricted weight-bearing and/or immobilization for at least one day
4. The patient reported a tendency to give way during functional activities
5. Positive anterior drawer test and/or talar tilt test
6. At least 2 giving-way episodes within 6 months before the study enrollment and/or recurrent ankle sprain
7. Score of 24 on the Cumberland ankle instability tool

Exclusion Criteria:

1. Acute ankle injuries within the past 3 months.
2. Any other lower extremity injuries or surgeries that could affect balance or ankle function.
3. Participation in either formal or informal rehabilitation before enrollment in the study
4. Skin allergy from kinesiotaping.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * fifty female athletes from will be recruited from the Faculty of Physical education for females, Helwan University.
  * Aged 18-24 years.
  * has a history of unilateral ankle inversion injury since at least one year before the study onset
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of Dorsiflexion range of motion | at baseline and after 2 weeks
  The weight-bearing lunge test is a controlled exercise that involves standing upright facing a vertical wall with a measuring tape and a tape affixed to the wall. Participants lunge forward, flexing at the ankle, knee, and hip on the test leg to make contact with the wall. After a successful attempt, the foot is moved backward in 1 cm increments. The distance between the heel and the wall and the anterosuperior edge of the patella is recorded to the nearest 0.1 cm. Ankle dorsiflexion angle is calculated using the trigonometric function.

SECONDARY OUTCOMES:
assessment of change of dynamic balance | at baseline and after 2 weeks
  The Y-balance test is a method to assess a person's dynamic balance by aiming to maintain single-leg balance while reaching as far as possible with the contralateral leg in three different directions. The test involves three trials for each reach direction, with resting intervals to minimize fatigue. To account for individual differences in limb length, reach distances are normalized to leg length. This method standardizes performance measurements, allowing for more accurate comparisons of dynamic balance and mobility between individuals of varying anthropometric characteristics. Normalization is essential in functional reach tasks to reduce bias and enhance the validity of inter-subject comparisons.
assessment of change of single-leg squat performance | at baseline and after 2 weeks
  The Kinovea software is used to assess single leg squat performance in patients with chronic ankle instability, focusing on stability and alignment. The patient's movements are captured using a high-resolution camera, ensuring clear view of lower extremities.
assessment of change of ankle physical function | at baseline and after 2 weeks
  The Foot and Ankle Ability Measure (FAAM) Sports Subscale is a tool used to measure physical function. It scores items from 4 to 0, with the highest potential score being the highest number of responses. Higher scores indicate better physical function, and the total score is divided by the highest potential score.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical education for females, Helwan university, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: No